CLINICAL TRIAL: NCT01291004
Title: A Multicenter, Open-Label Study to Evaluate Ovarian Follicular Activity and Hormone Levels With the Oral Contraceptive Regimen DR-102 Compared to Two 28-day Oral Contraceptive Regimens Containing Different Synthetic Progestins
Brief Title: A Study to Evaluate Ovarian Follicular Activity and Hormone Levels for DR-102 Compared to Two 28-Day Oral Contraceptives
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DSG-OI-101
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Follicle Development; Ovarian Follicle; Follicle Count; Follicle Size; Oral Contraceptive
MeSH Terms: interventions — Desogestrel; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 28-day Desogestrel Oral Contraceptive (Experimental)
  Interventions: Drug: Desogestrel/ethinyl estradiol and ethinyl estradiol
- 28-day Drospirenone Oral Contraceptive (Active Comparator)
  Interventions: Drug: 28-day drospirenone oral contraceptive
- 28-day Levonorgestrel Oral Contraceptive (Active Comparator)
  Interventions: Drug: 28-day levonorgestrel oral contraceptive

INTERVENTIONS:
Drug: Desogestrel/ethinyl estradiol and ethinyl estradiol — Desogestrel/ethinyl estradiol 0.15/0.02 mg and ethinyl estradiol 0.01 mg tablet
  Arms: 28-day Desogestrel Oral Contraceptive
Drug: 28-day drospirenone oral contraceptive — Drospirenone/ethinyl estradiol 0.3/0.02 mg
  Arms: 28-day Drospirenone Oral Contraceptive
Drug: 28-day levonorgestrel oral contraceptive — Levonorgestrel/ethinyl estradiol 0.1/0.02 mg
  Arms: 28-day Levonorgestrel Oral Contraceptive

SUMMARY:
This study is being conducted to evaluate the impact of a 28-day oral contraceptive compared to two 28-day oral contraceptive regimens containing different synthetic progestins on ovarian follicular activity and hormone levels in healthy women.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal, non-pregnant, non-lactating women age 18-35 years old
* Body Mass Index (BMI) ≥18 kg/m² and <30 kg/m²
* Regular spontaneous menstrual cycle
* Others as dictated by Food and Drug Administration (FDA)-approved protocol

Exclusion Criteria:

* Any condition which contraindicates the use of combination oral contraceptives
* Known thrombophlebitis or thromboembolic disorders; known or suspected clotting disorders; thrombogenic valvulopathies or rhythm disorders
* Migraine headaches with focal, neurological symptoms
* Others as dictated by FDA-approved protocol

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 206 (Actual)
Dates: Start 2011-01-31 (Actual); Primary Completion 2012-03-31 (Actual); Study Completion 2012-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of ovarian follicular development by the Hoogland and Skouby grading scale from baseline to week 16. | 16 weeks
Change in serum Estradiol level from baseline to week 16. | 16 weeks
Change in serum Follicle Stimulating Hormone (FSH) and Luteinizing Hormone (LH) levels from baseline to week 16. | 16 weeks
Change in serum Progesterone level from baseline to week 20. | 20 weeks

SECONDARY OUTCOMES:
Change from baseline to week 15 in Prothrombin fragment 1 + 2 levels. | 15 weeks
Change from baseline to week 15 in D-dimer. | 15 weeks
Change from baseline to end of week 15 in Plasmin-Antiplasmin complex | 15 weeks
Change from baseline to week 15 in APTT and ETP based activated protein-C resistance (APC). | 15 weeks
Change from baseline to week 15 in Fibrinogen. | 15 weeks
Change from baseline to week 15 in Plasminogen, Factor II, Factor VII, Factor VIII, Protein C, and Free and Total Protein S. | 15 weeks
Change from baseline to week 15 in Tissue Plasminogen Activator (t-PA). | 15 weeks
Change from baseline to week 15 in Antithrombin. | 15 weeks
Change from baseline to week 15 in Tissue Factor Pathway Inhibitor (TFPI). | 15 weeks
Change from baseline to week 15 in Total Cortisol and Corticosteroid Binding Globulin (CBG). | 15 weeks
Change from baseline to week 15 in Thyroid Stimulating Hormone (TSH). | 15 weeks
Change from baseline to week 15 in Sex Hormone Binding Globulin (SHBG). | 15 weeks
Return to ovulation rate at week 20. | Week 20

CONTACTS AND LOCATIONS:
Overall Officials: Teva Women's Health Research Protocol Chair, Study Chair — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (2):
- United States (2):
  - Teva Investigational Site 10119, Philadelphia, Pennsylvania
  - Teva Investigational Site 10118, Seattle, Washington